CLINICAL TRIAL: NCT06274034
Title: Pilot Study of a Wearable EEG Headband as a Meditation Device for Breast Cancer Survivors
Brief Title: MUSE-S Headband System for Improving Anxiety and Insomnia Among Breast Cancer Survivors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-006870; NCI-2024-01019 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-006870 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-02-15; First posted 2024-02-23 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (MUSE S headband, meditation) (Experimental): Patients wear the MUSE S headband to bed every night for 8 weeks and meditate using the MUSE phone app during day hours for at least 5 minutes over 8 weeks.
  Interventions: Other: Electronic Health Record Review; Other: Medical Device Usage and Evaluation; Procedure: Meditation Therapy; Other: Survey Administration

INTERVENTIONS:
Other: Electronic Health Record Review — Ancillary studies
Other: Medical Device Usage and Evaluation — Wear MUSE S headband
Procedure: Meditation Therapy — Participate in meditation
  Other Names: Meditation
Other: Survey Administration — Ancillary studies

SUMMARY:
This early phase I trial evaluates the feasibility and impact of a meditation headband system (MUSE-S) for breast cancer survivors. Anxiety and insomnia are among the most common distresses in breast cancer survivors during and after chemotherapy, in part due to the side effects of chemotherapy, fear of cancer coming back, progression of the cancer, and uncertainty of the future. These distresses impair patients' well-being and quality of life (QOL) in general, and their cancer treatment adherence and effectiveness in particular. Meditation has been demonstrated to be an effective management tool of stress and anxiety and is given the highest level of evidence (grade A) in the systematic review-based guidelines by the Society of Integrative Medicine. The portable, interactive, electroencephalographic (EEG) Muse headband guided meditation has been shown to improve fatigue, QOL, and stress in newly diagnosed breast cancer patients. The MUSE-S Headband System may decrease anxiety and insomnia among breast cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the frequency of use of meditation (a stress management technique) among breast cancer survivors.

II. To evaluate the feasibility of a wearable EEG headband, MUSE S, together with smartphone or tablet application (app) to guide breast cancer survivors' interactive meditation and sleep support.

III. To measure the impact of interactive meditation and sleep support through MUSE S among breast cancer survivors during or after chemotherapy on improving symptoms of anxiety and insomnia.

OUTLINE:

Patients wear the MUSE S headband to bed every night for 8 weeks and meditate using the MUSE phone app during day hours for at least 5 minutes over 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-80
* Breast cancer first diagnosed with stage 1-4 breast cancer in the past 10 years
* Patients report experiencing anxiety and insomnia both rated > 3 on a 0-10 scale (with 0 indicating none) at the time of enrollment
* Patients on anti-anxiety/anti-depressant medication must be on stable dose for 1 month prior to study enrollment and must stay on that same dose throughout the trial
* Has smart phone or tablet
* Patient willing to use Google-based anonymous email account to sign up for MUSE
* Be willing to provide informed consent and complete all aspects of the study
* Have no contraindicating comorbid health condition which would interfere with the proper use of the Muse-S (trademark) system, as determined by the clinical investigators

Exclusion Criteria:

* Pregnant or breastfeeding individuals
* Individuals who have used a regular mindfulness practice or received integrative medicine therapy, including acupuncture/acupressure, mindfulness or stress-reduction programs, massage, and/or energy therapies within the past 60 days
* Currently taking medication for insomnia
* An exclusionary unstable medical or mental health condition as determined by the patient's oncologist

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of use of meditation | Baseline; 6 weeks
  Assessed by the number of times participant uses the Muse™ S Headband system and app. Data will be downloaded from the Muse Dashboard to the study team.
Feasibility of a wearable electroencephalographic (EEG) headband (Muse™ S Headband) | 6 weeks
  Assessed by reviewing usage data and by post-study satisfaction questionnaire adapted from the Was it Worth it Questionnaire (WIWI) asking the patient if the entire research experience, including the intervention, was worth it for them. The WIWI questionnaire includes 3 items: (item 1) Was it worthwhile for you to receive the cancer treatment given in this study? (item 2) If you had to do it over again, would you choose to have this cancer treatment? and (item 3) Would you recommend this cancer treatment to others? Questions are answered with yes, uncertain, or no.
Impact of interactive meditation and sleep support through the Muse-S™ system | Baseline; 6 weeks
  Assessed by a 3-section questionnaire (sleep, quality of life, and anxiety) with a variety of questions answered by multiple choice (e.g., very well, somewhat well, not very well, not well at all) or answered on a scale of 1-10 where 1=as bad as it can band and 10=as good as it can be.

CONTACTS AND LOCATIONS:
Overall Officials: Stacy D. D'Andre, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials